CLINICAL TRIAL: NCT07281300
Title: Mindfulness-Oriented Respiratory Distress Symptom Intervention for Patients With Lung Cancer: A Feasibility Randomized Controlled Trial
Brief Title: Mindfulness-Oriented Respiratory Distress Symptom Intervention for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20250424001
Record Dates: First submitted 2025-06-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-05

CONDITIONS: Symptom Cluster; Breathlessness; Coughing; Fatigue Symptom; Lung Cancer Patients; Brain Activity
MeSH Terms: conditions — Syndrome; Dyspnea; Cough; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants cannot be blinded due to the nature of the intervention. However, they will be instructed to maintain confidentiality and avoid discussing intervention details with other participants to minimize potential biases. The outcomes assessor who collects the participant's information will be blinded to the group allocation. However, the statistician responsible for quantitative data analysis will work with de-identified and de-grouped datasets to ensure blinding during the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Oriented Respiratory Distress Symptom Intervention (M-RDSI) (Experimental): Patients in the M-RDSI group will receive a 6-week intervention, including 1) mindfulness training, such as mindful breathing and relaxation; 2) controlled breathing techniques, cough suppression techniques, acupressure, and exercise; and 3) using mindful breathing, relaxation, and attitudes to orientate the practice of RDSI.
  Interventions: Behavioral: Mindfulness-Oriented Respiratory Distress Symptom Intervention (M-RDSI)
- Usual care (Active Comparator): Usual care will receive health educational booklets and routine follow-ups offered by the oncology nurse in the cancer center that patients with lung cancer usually receive during the same 6 weeks.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Respiratory Distress Symptom Intervention (M-RDSI) — Patients in the M-RDSI group will receive a 6-week intervention and begin with a training session (ideally face-to-face at the cancer center or the research center or an online meeting as backup for around 60 minutes, including 1) mindfulness training, such as mindful breathing and relaxation; 2) controlled breathing techniques, cough suppression techniques, acupressure, and exercise; and 3) using mindful breathing, relaxation, and attitudes to orientate the practice of RDSI. A second group training session will be conducted 3 weeks later to review the intervention and discuss any questions participants may have. The training sessions will be delivered by a well-trained research assistant from experienced clinicians and the research team. Participants will be guided by the M-RDSI web-based educational materials (e.g., text, pictures, and videos) and a detailed intervention manual for their daily home practice.
  Arms: Mindfulness-Oriented Respiratory Distress Symptom Intervention (M-RDSI)
Other: Usual Care — Usual care will receive health educational booklets, including brief tips for symptom management designed by the research team, and routine follow-ups offered by the oncology nurse in the cancer center that patients with lung cancer usually receive.
  Arms: Usual care

SUMMARY:
Lung cancer is the leading cause of cancer mortality, posing a critical public health challenge in both Hong Kong and global populations. Patients with lung cancer frequently experience a distressing symptom cluster characterized by breathlessness-driven respiratory distress, accompanied by persistent cough and fatigue, which collectively impose a substantial disease burden. While our research team leader previously developed and validated a multi-component Respiratory Distress Symptom Intervention (RDSI) in England, demonstrating clinical efficacy for lung cancer management, its impact on psychological distress (anxiety and depression) proved limited. This limitation may reflect insufficient integration of psychological components, a crucial consideration given the well-established bidirectional relationship between respiratory symptoms and psychological distress. Emerging evidence indicates that mindfulness interventions provide dual therapeutic benefits by improving patient adherence and effectively addressing both physical symptoms, such as breathlessness and fatigue, as well as psychological distress, including anxiety and depression. Meanwhile, current evaluation methodologies have mainly focused on behavioral data collection, such as self-reported questionnaires, to reflect the effect before and after the intervention. Neuroimaging data can help understand the brain mechanisms underlying breathlessness and elucidate the effectiveness of interventions, thereby improving intervention strategies.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a mindfulness-oriented respiratory distress symptom intervention (M-RDSI) for patients with lung cancer. This study uses a two-phase experimental design to develop the M-RDSI and to evaluate the M-RDSI intervention's clinical and neurophysiological effects. In Phase I, the aim is to develop and content-validate the M-RDSI, including cultural adaptation adjustment and co-design of the M-RDSI intervention, including intervention teaching materials, through an expert panel consisting of patients with lung cancer and healthcare professionals. In Phase II, fifty participants will be randomized into the intervention group, receiving a 6-week M-RDSI intervention followed by a 12-week follow-up, or the control group, which will receive usual care during the same period. During Phase IIa, the feasibility, acceptability, and preliminary clinical outcomes will be evaluated. Feasibility will be assessed through recruitment, dropout, and retention rates. Acceptability will be measured by treatment adherence rates and participant satisfaction, gathered through qualitative interviews. Preliminary clinical effectiveness will include self-reported outcomes such as breathlessness, cough, fatigue, mindfulness, anxiety, depression, and quality of life. The generalized estimating equation will be employed to analyze the intervention effects. Additionally, one-on-one qualitative interviews will be conducted post-intervention to gather participants' feedback on the perceived effectiveness, acceptability, strengths, limitations, and suggestions for improving the M-RDSI program. In Phase IIb, a task-based fMRI will be conducted at baseline and post-intervention, using a set of breathlessness-related word cues as stimuli to assess changes in brain activity. Analysis will be corrected for multiple comparisons. A general linear model will be constructed for the first-level fMRI analysis. A 2-by-2 factorial ANOVA will assess the group-by-time interaction of brain activity, and a paired t-test will evaluate pre- and post-treatment changes within the intervention group for the group analysis.

ELIGIBILITY:
Inclusion Criteria:

* HK patients who can understand Cantonese, aged 18 years or older;
* A confirmed diagnosis of an intrathoracic malignancy, including small cell lung cancer, non-small cell lung cancer, or mesothelioma; at any stage of cancer treatment or palliative care;
* Self-reported impact on daily life from at least two of the three symptoms, where one symptom is breathlessness;
* Stability of COPD, if present;
* WHO Performance Status of 0-2;
* fMRI can be conducted;
* Expected lifespan of more than six months.

Exclusion Criteria:

* Cognitive impairments, severe psychotic symptoms, or other medical conditions that might hinder participation;
* Participating in mindfulness or other psychological support interventions or symptom management interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  The recruitment rate will be calculated as the percentage of eligible participants who enroll in the study out of the total number of eligible participants.
Retention rate | Immediately after intervention and at 12-weeks follow-up
  The retention rate will be calculated as the percentage of participants who completed the entire research process (including the follow-up) out of the initial recruitment number.
Drop-out rate | Immediately after intervention and at 12-weeks follow-up
  The drop-out rate will be calculated as the percentage of participants who voluntarily withdrew from the study out of the initial recruitment number.
Adherence rate | Immediately after intervention
  The adherence rate will be calculated as the percentage of participants who complete the 6-week intervention.
Participants' satisfaction | At 12-weeks follow-up
  The participants' satisfaction will be assessed through one-to-one interviews by well-trained PhD students or research assistants.

SECONDARY OUTCOMES:
Breathlessness | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Dyspnoea-12. Participants will be asked to rate 12 items, with each item scored on a scale from 0 to 3. The total score ranges from 0 to 36, with higher scores indicating more severe symptoms of breathlessness.
Breathlessness expectation | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Breathlessness word cue set. Participants will be asked to rate 23 items using two Visual Analogue Scales: one for breathlessness and the other for breathlessness-anxiety. Each item ranges from 0% to 100%, with higher scores indicating greater levels of breathlessness or breathlessness-anxiety.
Cough | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Leicester Cough Questionnaire. Participants will be asked to rate 19 items, each scored on a scale from 1 to 7. The total score is calculated by converting the item scores, yielding a possible range from 3 to 21, with higher scores indicating less severe cough symptoms.
Fatigue | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Functional Assessment of Chronic Illness Therapy-Fatigue. Participants will be asked to rate 13 items, each scored on a five-point Likert scale from 0 to 4. The total score ranges from 0 to 52, with higher scores indicating less severe fatigue symptoms.
Mindfulness | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Mindful Attention Awareness Scale. Participants will be asked to rate 15 items, each scored on a six-point Likert scale from 1 to 6. The overall score is obtained by averaging the scores of all items, with higher mean scores indicating a greater level of mindfulness.
Depression | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the Center for Epidemiologic Studies Depression Scale. Participants will be asked to rate 20 items, each scored on a four-point Likert scale from 0 to 3. The total score ranges from 0 to 60, with higher scores indicating more severe depressive symptoms.
Anxiety | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the State-Trait Anxiety Inventory, which consists of two subscales: the State Anxiety Scale and the Trait Anxiety Scale. Each subscale contains 20 items, with each item scored on a four-point Likert scale from 1 to 4. The total score for each subscale ranges from 20 to 80, with higher scores indicating greater levels of state or trait anxiety.
Quality of life (QoL) | Baseline, immediately after intervention, and at 12-weeks follow-up
  This will be measured by the EuroQoL 5-Dimension 5-Level. Participants will be asked to rate five domains-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each on a five-level scale ranging from no problems to extreme problems. Participants will also be asked to provide an overall assessment of their health using a visual analogue scale from 0 to 100, with higher visual analogue scale scores indicating better quality of life.
Breathlessness expectation-related brain activity | Baseline and immediately after intervention.
  A task-based fMRI technology will be used to measure breathlessness expectation using a breathlessness word cue set.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No